CLINICAL TRIAL: NCT04645732
Title: Improving Health in People With Multimorbidity: a Paradigm Shift in Health Care From Disease-based Curative Models to Personalized Exercise Therapy and Self-management
Brief Title: Personalized Exercise Therapy and Self-management Support for Patients With Multimorbidity
Acronym: MOBILIZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Naestved Hospital (Other); Slagelse Hospital (Other); Lolland Municipality (Unknown); Roskilde Municipality (Unknown); Psychiatric Hospital West, Slagelse (Unknown); Næstved, Slagelse and Ringsted Hospitals' Research Fund (Unknown); Association of Danish Physiotherapists (Other); The Danish Health Confederation through the Development and Research Fund (Unknown); European Research Council (Other); Holbaek Sygehus (Other); Nykøbing Falster County Hospital (Other); FysioDanmark Holbæk (Unknown); Zealand University Hospital (Other); Lægerne Reventlow og Wolfhagen, Slagelse (Unknown); Lægerne Algade 17, Roskilde (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJ-857; 801790 (Other Grant/Funding Number: European Research Council under the EU Horizon 2020 program)
Record Dates: First submitted 2020-11-02; First posted 2020-11-27 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Heart Failure; Coronary Heart Disease; Hypertension; Type2 Diabetes; Chronic Obstructive Pulmonary Disease; Depression
Keywords: Exercise; Self-management; Clinical Trial; Multimorbidity; Evaluation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Heart Failure; Coronary Disease; Hypertension; Pulmonary Disease, Chronic Obstructive; Depression; Motor Activity

STUDY DESIGN:
Intervention Model Description: The RCT is a pragmatic, parallel-group, superiority RCT (1:1 ratio)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study investigators, outcome assessors and the statistician will be blinded to randomization. Furthermore, a blinded interpretation of the study results will be conducted
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized exercise therapy and self-management program in addition to usual care (Experimental): Participants randomized to the personalized exercise therapy and self-management support program will participate in a 12-week program tailored to people with multimorbidity at one of the intervention sites. The program will consist of 24 exercise therapy and self-management sessions distributed across the program (twice weekly, each lasting around 1.5 hour).
  Furthermore, this group will receive the treatment described under usual care below.
  Interventions: Behavioral: Personalized exercise therapy and self-management support program; Other: Usual care
- Usual care alone (Active Comparator): Usual care is the care that the participants would receive had they not participated in the study, i.e. treatments or services that are routinely provided in the settings from which the participants are recruited. Participants will continue their current treatment, if needed, and be allowed to receive other treatments if their general practitioner or specialist finds it relevant for their particular comorbidities.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Personalized exercise therapy and self-management support program — See description under Arms
  Arms: Personalized exercise therapy and self-management program in addition to usual care
Other: Usual care — See description under Arms

SUMMARY:
Chronic conditions such as knee or hip osteoarthritis (OA), chronic obstructive pulmonary disease (COPD), heart failure (HF), coronary heart disease (CHD), hypertension, type 2 diabetes mellitus (T2DM) and depression are among the leading causes of global disability and affect hundreds of millions of people around the world. In recent years, multimorbidity, commonly defined as the co-occurrence of at least two chronic conditions, has also gained interest due to its substantial impact on the person and society.

Despite the significant burden of multimorbidity, little is known about how to treat this effectively. A 2016 Cochrane systematic review found that interventions targeting populations with specific combinations of conditions and addressing specific problems such as functional difficulties may be more effective. Exercise therapy is a treatment addressing functional limitations that is a safe and effective treatment of at least 26 chronic conditions, including OA, HF, CHD, hypertension, T2DM, COPD and depression. Furthermore, self-management support is increasingly recognized as an essential component of interventions to improve outcomes in patients living with multimorbidity and to support the long-term adherence to exercise. A new systematic review found that exercise seems effective in people with multimorbidity (the conditions included in the current study), however highlighting the need for further high-quality RCTs.

The aim of this randomized controlled trial (RCT) is to investigate the effects of a personalized exercise therapy and self-management support program in addition to usual care on self-reported, objectively measured and physiological outcomes in people with multimorbidity (i.e. at least two of the following conditions: OA (knee or hip), heart condition (HF or CHD), hypertension, T2DM, COPD and depression). The primary endpoint is 12 months, but 4- and 6-month follow-ups are included as well and a 12-month health economic evaluation of the program will be conducted.

Prior to the RCT, a feasibility trial of 20 people with multimorbidity, all undergoing the personalized exercise therapy and self-management support program, will be conducted using the same methods as in the RCT, but primarily focusing on feasibility outcomes (recruitment, retention, adherence to treatment, burden of outcomes, improvements in outcomes, adverse events). This will start recruitment in Feb 2021 and end August 2021.

The MOBILIZE project has received funding from several foundations, including the European Research Council (ERC) under the European Union's Horizon 2020 research and innovation program (grant agreement No 801790).

DETAILED DESCRIPTION:
Chronic conditions such as knee or hip osteoarthritis (OA), chronic obstructive pulmonary disease (COPD), heart failure (HF), coronary heart disease (CHD), hypertension, type 2 diabetes mellitus (T2DM) and depression are among the leading causes of global disability and affect hundreds of millions of people around the world. In recent years, multimorbidity, commonly defined as the co-occurrence of at least two chronic conditions, has also gained interest due to its substantial impact on the person and society. In general, multimorbidity affects more than half of all people with chronic conditions. Two out of three people with OA have comorbidities, with HF, CHD, hypertension, T2DM, COPD and depression being some of the most common.

People with multimorbidity account for 78% of all consultations in primary care and multimorbidity is associated with poorer function and quality of life, depression, intake of multiple drugs and increased health care utilization, with some studies demonstrating an almost exponential relationship between the number of chronic conditions and their health care costs. Furthermore, we know from qualitative research that treating one condition at a time is inconvenient, inefficient and unsatisfactory for the person with the chronic conditions and his or her health care provider. Most research so far has excluded people with multimorbidity, due to its focus on only one specific condition, and most of the health care sector manages each individual condition on its own instead of the person, highlighting the negative impact of the current disease-based curative models on multimorbidity. With a population that is ageing, and a significant number of people with multimorbidity being younger than 65 years of age, the proportion of people with multimorbidity is increasing rapidly, emphasizing the need to take action to deal with the increasing burden of chronic conditions and multimorbidity through treatment and prevention.

Identifying and developing effective and affordable treatment strategies to deal with the global burden of chronic conditions and multimorbidity is a major focus of modern health care around the world. Despite the significant burden of multimorbidity, little is known about how to treat this effectively. A 2016 Cochrane systematic review found that interventions targeting populations with specific combinations of conditions and addressing specific problems such as functional difficulties may be more effective. A treatment addressing functional limitations that is able to improve symptoms in at least 26 chronic conditions, including OA, HF, CHD, hypertension, T2DM, COPD and depression is readily available. This treatment is exercise therapy, which is effective, safe and supported by substantial evidence in patients with knee and hip OA, HF and CHD, hypertension, T2DM, COPD, depression and a range of other chronic conditions. A new systematic review found that exercise seems effective in people with multimorbidity (the conditions included in the current study), however highlighting the need for further high-quality RCTs. Furthermore, self-management support is increasingly recognized as an essential component of interventions to improve outcomes in patients living with multimorbidity. There is increasing evidence that effective management of multimorbidity requires the active participation by patients in the care process. Self-management support interventions have been shown to change health behaviors, improve health status, and reduce health care utilization and costs. Self-management support is centered on enabling patients to develop a set of behavioral skills and abilities to help them navigate a range of disease management tasks across different chronic conditions.

In an RCT of people with knee OA, published in the New England Journal of Medicine, we found that 3 out of 4 patients eligible for total knee replacement improved enough from self-management support, supervised exercise therapy and other non-surgical treatments to postpone surgery for at least one year. Furthermore, in patients with T2DM, 56% did not take antidiabetic medication after 1 year of supervised exercise therapy, self-management support and diet. Together, these studies indicate the potential of combining exercise, self-management and other treatments to reduce the need for surgery and medication. A recent cohort study found that an eight-week exercise and self-management program demonstrated similar improvements in health outcomes for people with OA and the comorbidities included in the current study as for people without comorbidities.

Altogether, this highlights exercise therapy and self-management support as viable treatment options for people with multimorbidity, but the evidence supporting this is of low quality and more high-quality RCTs are needed to improve care for the millions of people suffering from multimorbidity worldwide.

The overall aim of the MOBILIZE project is to empower patients with multimorbidity to take a more active role in their health care through a personalized exercise therapy and self-management support program so that they may reduce symptoms of the individual conditions, increase quality of life and physical function and prevent development of other chronic conditions. To ensure relevance to the patients and the health care system and to make sure that the project is implementable in clinical practice afterwards, strong interdisciplinary collaboration involving many different scientific methodologies and a high degree of patient involvement throughout the entire research process are at the heart of the project. The MOBILIZE project has received funding from several foundations, including the European Research Council (ERC) under the European Union's Horizon 2020 research and innovation program (grant agreement No 801790). Building on the Medical Research Council's framework for the development and evaluation of complex interventions, the MOBILIZE project has four phases. During the first phase of the project, outcomes and biomarkers that predict better health outcome from different types of exercise therapy and exercise characteristics associated with a better outcome in people with different combinations of chronic conditions will be identified through exploratory observational cohort studies of people with osteoarthritis who have undergone an 8-week exercise therapy and education program in Denmark (GLA:D) as well as scoping reviews, systematic reviews and meta-analyses that summarize the existing evidence. Subsequently, in phase 2, a 12-week exercise therapy and self-management support program will be developed based on existing recommendations for exercise and strategies to facilitate behavioral changes. To ensure a high degree of patient and provider involvement, focus group interviews will be conducted with patients with multimorbidity, health care providers and other relevant stakeholders to acquire their views and perspectives on multimorbidity and exercise. Once this phase is completed, the exercise therapy and self-management support program will be tested in a feasibility trial involving 20 patients with multimorbidity (recruited from Feb 2021 and onwards). The same procedures and outcomes as in the subsequent RCT will be used, and data will be collected at baseline and after the 12-week intervention. The feasibility trial will primarily focus on feasibility outcomes (recruitment, retention, adherence to treatment, burden of outcomes, improvements in outcomes, adverse events), using a red/amber/green traffic light system, guiding the progression to the subsequent RCT. Experiences from the feasibility trial will be used to evaluate and implement any adjustments that need to be made prior to commencing the RCT (described in details in the current trial registration). The RCT corresponds to phase 3, while phase 4 focuses on developing a model for implementation of the personalized exercise therapy and self-management support program in clinical practice, if supported by the study findings.

The aim of the RCT described in this clinical trial registration is to investigate the effects of a personalized exercise therapy and self-management support program in addition to usual care on self-reported, objectively measured and physiological outcomes in people with multimorbidity (i.e. at least two of the following conditions: OA (knee or hip), heart condition (HF or CHD), hypertension, T2DM, COPD and depression). The primary endpoint is 12 months, but 4- and 6-month follow-ups are included as well and a 12-month health economic evaluation of the program will be conducted. The 4-month follow-up corresponds to immediately after the intervention, including the time it takes to conduct the baseline measurements and be enrolled in the group-based program.

The primary study hypothesis is that a personalized exercise therapy and self-management support program in addition to usual care will improve quality of life more than usual care alone when measured at 12 months with concurrent positive effects on secondary outcomes. Furthermore, it is hypothesized that the program will be cost-effective at 12 months.

People will be recruited via the recruitment centers mentioned in this registration as well as via self-referral (Facebook posts, newspaper articles and flyers).

People who only fulfil some of the eligibility criteria (aged 18 years or above, at least two of the relevant conditions and do not have psychosis disorders, post-traumatic stress disorder, Obsessive Compulsive Disorder, attention deficit hyperactivity disorder, autism, anorexia nervosa/bulimia nervosa or an abuse or other reasons for exclusion) or people fulfilling all eligibility criteria, but unwilling to participate in the RCT, will be offered participation in an observational cohort study where only the self-reported outcomes are completed. Recruitment for the cohort will start and end with the recruitment for the RCT.

ELIGIBILITY:
Inclusion Criteria:

* At least two of the following conditions: OA (knee or hip), COPD, heart condition (HF or CHD), hypertension, T2DM, depression (having other comorbidities does not exclude a patient)
* Adults aged 18 years or above
* Able to walk 3 meters without any assistance
* A score of 3 or above on the Bayliss' Disease Burden: Morbidity Assessment by Self- Report scale for at least one of the conditions listed above and a score of 2 or above for at least one of the other listed conditions
* Willingness and ability to participate in a 12-week supervised exercise therapy and self- management support program twice a week

Exclusion Criteria:

* Participation in supervised systematic exercise for one of their diseases within the last 3 months
* Patients with an unstable health condition or at risk of serious adverse events as evaluated by a medical specialist
* Patients categorized as Class IV on the New York Heart Association (NYHA) Functional Classification scale
* Terminal patients and patients with life expectancy of less than 12 months
* Patients with psychosis disorders, post-traumatic stress disorder, Obsessive Compulsive Disorder, attention deficit hyperactivity disorder, autism, anorexia nervosa/bulimia nervosa and patients with dependency disorders
* Other reasons (unable to understand Danish, mentally unable to participate, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
EQ-5D-5L, the descriptive index | Primary endpoint: Change from baseline to 12 months
  The descriptive index of the EuroQol-5 Domain 5-level questionnaire (EQ-5D-5L) measures the patient's self-rated health status. Ranging from -0.757 to 1, higher is better. This will also allow for a later cost-effectiveness analysis. Assessed at baseline, 4, 6 and 12 months. All visits (baseline, 4, 6 and 12 months) will be included in the analysis.

SECONDARY OUTCOMES:
6-minute walk test | Primary endpoint: Change from baseline to 12 months
  The walking distance covered over a time of 6 minutes. Assessed at baseline, 4 and 12 months.
Burden of illness measure | Primary endpoint: Change from baseline to 12 months
  The burden of illness measure developed by Bayliss et al. measures how much illness affects the individual's daily activities (on a 1-5 scale for each individual condition, higher is worse, summed to a total score for all conditions, with an upper limit depending on the number of conditions included). Assessed at baseline, 4, 6 and 12 months.
30-second chair-stand test | Primary endpoint: Change from baseline to 12 months
  The number of chair stands completed in 30 seconds. Assessed at baseline, 4 and 12 months.
Depression Scale | Primary endpoint: Change from baseline to 12 months
  Personal Health Questionnaire Depression Scale (PHQ-8). Ranging from 0-24 points, higher is more severe depression. Assessed at baseline, 4, 6 and 12 months.
Anxiety | Primary endpoint: Change from baseline to 12 months
  General Anxiety Disorder-7 (GAD-7). Ranging from 0-21, higher is more severe anxiety. Assessed at baseline, 4, 6 and 12 months.
Self-Efficacy | Primary endpoint: Change from baseline to 12 months
  Self-Efficacy for Managing Chronic Disease 6-item Scale. Mean of 6 items, ranging from 1 to 10, higher scores indicating higher self-efficacy. Assessed at baseline, 4, 6 and 12 months.
Overall functioning and disability | Primary endpoint: Change from baseline to 12 months
  12-item WHO Disability Assessment Schedule 2.0 (WHODAS 2.0). Ranging from 0 (no disability) to 100 (full disability). Assessed at baseline, 4, 6 and 12 months.
Adverse events | Primary endpoint: 12 months
  Adverse events (AE) and serious adverse events (SAE) will be recorded at all follow-ups by asking the participants about potential AEs using open-probe questioning to ensure that all AEs are recorded. Furthermore, the medical records of the patients will be checked at the primary endpoint (12 months) for all AEs occurring from inclusion until the 12 months follow-up. AEs will be classified according to the Food and Drug Administration definition of an SAE and recorded, categorized and assessed for severity independent of whether or not there is a causal relationship with study treatments. Assessed at 4, 6 and 12 months.
Steps per day | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
Minutes/day spent being physically active with at least light intensity | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
EQ-5D-5L, the subscale EQ VAS | Primary endpoint: Change from baseline to 12 months
  The EQ visual analogue scale (EQ VAS) evaluates the patient's self-rated health on a 0-100 vertical visual analogue scale, higher score is better. Assessed at baseline, 4, 6 and 12 months.
Mortality | Primary endpoint: 12 months
  Mortality will be recorded at 12 months via medical records

OTHER OUTCOMES:
Isometric knee-extension strength | Primary endpoint: Change from baseline to 12 months
  Isometric knee-extension strength assessed using a hand-held dynamometer. Assessed at baseline, 4 and 12 months.
Balance | Primary endpoint: Change from baseline to 12 months
  Tandem 30-second balance test. Assessing balance in 30-second with 10 seconds in each of the 3 different positions (parallel feet, semi-tandem and tandem stand) resulting in a score from 0-30, higher is better. Assessed at baseline, 4 and 12 months.
Pain (yes/no) in left and right knee and hip + worst joint if more than one | Primary endpoint: Change from baseline to 12 months
  Left/right knee/hip pain + worst joint if more than one. Assessed at baseline, 4, 6 and 12 months.
Stress | Primary endpoint: Change from baseline to 12 months
  Perceived Stress Scale (4-item version). Ranging from 0-16, higher is more stressed. Assessed at baseline, 4, 6 and 12 months.
Systolic and diastolic blood pressure | Primary endpoint: Change from baseline to 12 months
  Blood pressure after 5 minutes of rest. Assessed at baseline, 4 and 12 months.
Concentration of cholesterol (HDL and LDL) and triglyceride | Primary endpoint: Change from baseline to 4 months
  Levels of cholesterol (HDL and LDL) and triglyceride. Assessed at baseline and 4 months.
Concentration of Fasting glucose | Primary endpoint: Change from baseline to 4 months
  Levels of fasting glucose. Assessed at baseline and 4 months.
Concentration of Fasting insulin | Primary endpoint: Change from baseline to 4 months
  Levels of fasting insulin. Assessed at baseline and 4 months.
Concentration of HbA1c | Primary endpoint: Change from baseline to 4 months
  Levels of HbA1c. Assessed at baseline and 4 months.
Concentration of high-sensitivity C-reactive protein (hs-CRP) | Primary endpoint: Change from baseline to 4 months
  Levels of the inflammatory marker high-sensitivity C-reactive protein (hs-CRP). Assessed at baseline and 4 months.
Concentration of Tumor necrosis factor (TNF) | Primary endpoint: Change from baseline to 4 months
  Levels of the inflammatory marker Tumor necrosis factor (TNF). Assessed at baseline and 4 months.
Concentration of Interleukin 6 (IL-6) | Primary endpoint: Change from baseline to 4 months
  Levels of the inflammatory marker Interleukin 6 (IL-6). Assessed at baseline and 4 months.
Concentration of Interleukin-1 receptor antagonist (IL-1ra) | Primary endpoint: Change from baseline to 4 months
  Levels of the inflammatory marker Interleukin-1 receptor antagonist (IL-1ra). Assessed at baseline and 4 months.
Weight | Primary endpoint: Change from baseline to 12 months
  Weight in kg. measured with a scale. Assessed at baseline, 4 and 12 months.
Adapted Fried Frailty and pre-frailty criteria | Primary endpoint: Change from baseline to 12 months
  Frailty and pre-frailty assessed by the Adapted Fried Frailty and pre-frailty criteria. Assessed at baseline, 4 and 12 months.
Fatigue | Primary endpoint: Change from baseline to 12 months
  One-item self-reported fatigue. Assessed at baseline, 4, 6 and 12 months.
Disease-specific treatment | Primary endpoint: Change from baseline to 12 months
  Self-reported disease-specific treatment. Assessed at baseline, 4, 6 and 12 months.
Knee/hip pain, VAS | Primary endpoint: Change from baseline to 12 months
  Average knee/hip pain during the last 7 days on a 0-100 visual analogue scale for worst joint (higher is worse pain, only for patients reporting knee/hip pain). Assessed at baseline, 4, 6 and 12 months.
Patient Acceptable Symptom State (PASS) | Primary endpoint: 12 months
  "Thinking about your quality of life, would you consider your current health as satisfying? With quality of life, you should consider your activities of daily living, sport and recreational activities, personal care, level of pain, and any anxiety or depression." Answered by "yes" or "no". Assessed at 4, 6 and 12 months.
Patient-reported treatment failure | Primary endpoint: 12 months.
  Only answered by patients answering "no" to PASS. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?". Answered by "yes" or "no". Assessed at 4 and 12 months.
Adherence | Primary endpoint: 4 months
  Adherence to intervention protocol of the study assessed as the number of exercise and self-management support sessions attended out of the total number of sessions available. Assessed at 4 months.
Other treatment during follow-up | Primary endpoint: 12 months
  Assessed by asking the patient about changes in their pharmacological treatment as well as any other treatments that they have received outside the study since the last assessment. If the patient answers yes, questions on details of the changes and other treatments will be asked. Assessed at 4, 6 and 12 months.
Work status | 12 months.
  "What is your current work status?" The patients choose one of several categories (e.g. "Working", "On sick leave, full time" and "Pensioner". Assessed at baseline, 4, 6 and 12 months.
Smoking | Primary endpoint: 12 months
  "How many cigarettes did you smoke in the last 7 days?" Assessed at baseline, 4, 6 and 12 months.
Questionnaire burden (only feasibility study) | Primary endpoint: 4 months
  "Did you find the questionnaire so burdensome that you would not participate in the study again?" Answered "yes"/"no". Assessed at baseline and 4 months.
Assessment burden (only feasibility study) | Primary endpoint: 4 months
  "Did you find the assessments so burdensome that you would not participate in the study again?" Answered "yes"/"no". Assessed at baseline and 4 months.
Isometric handgrip strength | Primary endpoint: Change from baseline to 12 months
  Isometric handgrip strength assessed using a hand-held dynamometer. Assessed at baseline, 4 and 12 months.
Multimorbidity Treatment Burden | Primary endpoint: Change from baseline to 12 months
  Multimorbidity Treatment Burden Questionnaire. Ranging from 0-100, higher is worse. Assessed at baseline, 4, 6 and 12 months.
Short form of Patient Activation Measure (PAM) | Primary endpoint: Change from baseline to 12 months
  Short form of Patient Activation Measure (PAM). Ranging from 0-100, higher scores indicating higher levels of patient activation. Assessed at baseline, 4, 6 and 12 months.
Bodily pain | Primary endpoint: Change from baseline to 12 months
  The number of self-reported body sites with pain in the previous 24 hours reported on a region-divided body chart of the front (A) and back (B) sides of the body. Assessed at baseline, 4, 6 and 12 months.
Sedentary behaviour | Primary endpoint: Change from baseline to 12 months
  Daily sedentary behaviour (one item). Assessed at baseline, 4, 6 and 12 months.
Individual items from the 12-item WHODAS 2.0 | Primary endpoint: Change from baseline to 12 months
  The 12 individual items from WHO Disability Assessment Schedule 2.0. Ranging from 1 to 5, higher score is worse. Assessed at baseline, 4, 6 and 12 months.
Spirometry (FEV1) | Only assessed at baseline.
  Spirometry (MedikroPro) will be used to measure forced expiratory volume in first second in liter (FEV1).Assessed at baseline.
Self-reported physical activity level | Primary endpoint: Change from baseline to 12 months
  Weekly physical activity (two items). Assessed at baseline, 4, 6 and 12 months.
Global Perceived Effect (GPE) | Primary endpoint: 12 months
  Global Perceived Effect (GPE) for physical activity level, activities of daily living and quality of life. Answered on 7-point Likert scale ranging from (1) "Much better, an important improvement" to (7) "Much worse, an important deterioration", higher score is worse. Assessed at 4, 6 and 12 months.
Falls | Primary endpoint: 12 months
  Over the last 4 months, have you ever been falling? "2months" at 6-month follow-up and "6 months" at the 12-month follow-up. (A fall is defined as an event resulting in you inadvertently coming to rest on the ground or another lower level, with or without loss of consciousness or injury). Never; Once; Twice; Three times or more. Assessed at 4, 6 and 12 months.
Fear of falling | Primary endpoint: 12 months
  How concerned are you that you might fall? Not at all concerned; Somewhat concerned, Fairly concerned, Very concerned. Assessed at 4, 6 and 12 months.
Sedentary activity: Time spent on sedentary activities | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
Light physical activity: Time spent on light intensity activities | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
Moderate physical activity: Time spent on moderate intensity activities | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
Vigorous physical activity: Time spent on vigorous intensity activities | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
Moderate to vigorous physical activity: Time spent on moderate to vigorous intensity activities | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
Adherence to the World Health Organization (WHO) physical activity recommendations, i.e. ≥150 min. MVPA or ≥75 min. VPA weekly activities | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
Sleep, objectively measured | Primary endpoint: Change from baseline to 12 months
  Objectively measured sleep assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
Sleep quantity, self-reported | Primary endpoint: Change from baseline to 12 months
  Self-reported average sleep quantity. Assessed at baseline, 4, 6 and 12 months.
Modified Karolinska Sleep Questionnaire | Primary endpoint: Change from baseline to 12 months
  Sleep quality will be measured by the Modified Karolinska Sleep Questionnaire (4 items). Ranging from 4 to 24, lower is worse sleep quality. Assessed at baseline, 4, 6 and 12 months.
Vigorous Intermittent Lifestyle Physical Activity (VILPA). | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.
Moderate-to-Vigorous Intermittent Lifestyle Physical Activity (MV-ILPA). | Primary endpoint: Change from baseline to 12 months
  Objectively measured physical activity assessed using combined wearable thigh and wrist accelerometers. Assessed at baseline, 4 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Søren T Skou, PT, MSc, PhD, Principal Investigator — Næstved, Slagelse and Ringsted hospital and University of Southern Denmark; Uffe Bødtger, MD, Study Chair — Department of Pulmonology, Næstved Hospital; Peter Gæde, MD, Study Chair — Department of Cardiology and Endocrinology, Slagelse Hospital; Manuel J Bieder, MD, Study Chair — Department of Orthopaedic Surgery, Næstved Hospital; Sidse Arnfred, MD, Study Chair — Psychiatric Hospital West, Slagelse; Christine Bodilsen, PT, MSc, PhD, Study Chair — Municipality of Roskilde; Jan A Overgaard, PT, MSc, Study Chair — Municipality of Lolland; Alessio Bricca, MSc, PhD, Study Chair — Næstved, Slagelse and Ringsted hospital and University of Southern Denmark; Madalina Jäger, MSc, PhD, Study Chair — Næstved, Slagelse and Ringsted hospital and University of Southern Denmark; Christian S Christiansen, MD, Study Chair — Nykøbing Falster County Hospital; Anne Merete B Soja, MD, PhD, DMSc, Study Chair — Holbaek Sygehus; Niels Eske Bruun, MD, Study Chair — Department of Cardiology, Zealand University Hospital, Roskilde; Johan L Reventlow, MD, Study Chair — Lægerne Reventlow og Wolfhagen, Slagelse; Andreas Heltberg, MD, PhD, Study Chair — Lægerne Algade 17, Roskilde; Lau C Thygesen, MSc, PhD, Study Chair — University of Southern Denmark; Poul Erik Holst, MD, Study Chair — Læge Poul Erik Holst, Holbæk; Rita M Andersen, MSc, Study Chair — Psychiatric Clinic Næstved; Amir Pasha Attarzadeh, MD, Study Chair — Department of Orthopedics, Zealand University Hospital, Køge; Mickey T Kongerslev, MSc, Study Chair — Community Psychiatry Roskilde; Louise Richelieu, MD, Study Chair — Lægehuset Tolskovvej, Hvalsø; Signe Aspelin, MD, Study Chair — Lægehuset Ostenfeldt, Næstved; Sille Capion, MD, Study Chair — Lægehuset Ostenfeldt, Næstved; Rune F Nielsen, Nurse, Study Chair — Community Clinic Nakskov
Locations (16):
- Denmark (16):
  - Holbæk Sygehus, Holbæk
  - Læge Poul Erik Holst, Holbæk
  - Lægehuset Tolskovvej, Kirke Hvalsø
  - Department of Orthopedics, Zealand University Hospital, Køge
  - Community Clinic, Nakskov
  - Department of Orthopaedic Surgery, Næstved Hospital, Næstved
  - Department of Pulmonology, Næstved Hospital, Næstved
  - Lægehuset Ostenfeldt, Næstved
  - Psychiatric Clinic Næstved, Næstved
  - Community Psychiatry Roskilde, Roskilde
  - Department of Cardiology, Zealand University Hospital, Roskilde
  - Lægerne Algade 17, Roskilde
  - Department of Cardiology and Endocrinology, Slagelse Hospital, Slagelse
  - Lægerne Reventlow og Wolfhagen, Slagelse
  - Psychiatric Hospital West, Slagelse, Slagelse
  - Nykøbing Falster County Hospital, Slagelse

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request after the primary publications have been published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Ultimo 2024.
Access Criteria: Data will be made available upon reasonable request after the primary publications have been published.
URL: https://osf.io/qk6yg/

REFERENCES:
- [Derived] Skou ST, Nyberg M, Dideriksen M, Rasmussen H, Overgaard JA, Bodilsen C, Soja AMB, Attarzadeh AP, Bieder MJ, Dridi NP, Heltberg A, Gaede PH, Reventlow JL, Arnfred S, Bodtger U, Brond JC, Thygesen LC, Moller SP, Jager M, Bricca A. Exercise therapy and self-management support for individuals with multimorbidity: a randomized and controlled trial. Nat Med. 2025 Sep;31(9):3176-3182. doi: 10.1038/s41591-025-03779-4. Epub 2025 Jun 30. PMID 40588675
- [Derived] Skou ST, Brodsgaard RH, Nyberg M, Dideriksen M, Bodtger U, Bricca A, Jager M. Personalised exercise therapy and self-management support for people with multimorbidity: feasibility of the MOBILIZE intervention. Pilot Feasibility Stud. 2023 Jan 18;9(1):12. doi: 10.1186/s40814-023-01242-0. PMID 36653858
- See also: Open Science Framework platform for MOBILIZE — https://osf.io/qk6yg/
- See also: MOBILIZE webpage — https://www.mobilize-project.dk/?lang=en